CLINICAL TRIAL: NCT06142929
Title: Observational Study on Small Nerve Bundles in Dupuytren Disease and the Impact of Its Dissection on Recurrence.
Brief Title: Micronerves in Dupuytren and the Impact of Its Dissection on Recurrence
Acronym: Micronerves
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68137
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Dupuytren disease: 50 patients with primary Dupuytren disease that are selected for surgery and will undergo the resection of Dupuytren tissue with the microfasciectomy technique
  Interventions: Procedure: Microfasciectomy
- Recurrence Dupuytren disease: 30 patients with recurrence Dupuytren disease that are selected for surgery and will undergo the resection of Dupuytren tissue with the microfasciectomy technique
  Interventions: Procedure: Microfasciectomy

INTERVENTIONS:
Procedure: Microfasciectomy — Using the microscope in Dupuytren's surgery

SUMMARY:
Dupuytren disease (DD) is a highly prevalent disabling hand disease. Spontaneous fibrosis nodules and strands in the palms of the hand cause finger contractures in disturbing positions and movement restrictions. Finger movement can be restored by surgery (removing the fibrosis tissue), but recurrence is a major problem and this is difficult to treat.

Through microfasciectomy, the presence of small nerve bundles (micronerves) were observed. These nerves are possibly related to the hand fascia, which is the origin of Dupuytren disease. These micornerves and their dissection could play a role in the recurrence of DD. This study will investigate the role of these micronerves in DD, the impact of its dissection on formation of neuromas and on recurrence.

Also, the presence of nerve growth factor (NGF) will be evaluated. The purpose is to provide information on potential neuro-induced fibrosis.

DETAILED DESCRIPTION:
Dupuytren disease (DD) is a highly prevalent disabling hand disease. Spontaneous fibrosis nodules and strands in the palms of the hand cause finger contractures in disturbing positions and movement restricitions. Finger movement can be restored by surgery (removing the fibrosis tissue), but recurrence is a major problem (reports of >70%) and this is difficult to treat.

Through microfasciectomy, the presence of small nerve bundles (micronerves) were observed in the finger (other than the digital nerves) through microsurgical enlargement. These nerves are possibly related to the hand fascia, which is the origin of DD. Palmaris fascia innervation was recently elucidated in 16 cadavers and recent research had demonstrated that the palmar aponeurosis is densely innervated and contains a variety of sensory corpuscles as wall as free nerve endings.

These micronerves and their dissection could play a role in the recurrence of DD. This thought is substantiated by the fact neuromas (formed by transection of nerves) were found in recurrence DD and nerve damage is generally known to cause fibrosis (as seen in chronic reactive pain syndrome). This study will investigate the role of these micronerves in DD, the impact of its dissection on formation of neuromas and on recurrence.

It's an observational study, investigation 2 groups of patients. Group 1 being patients with primary DD and group 2 patients with recurrence DD. The nerves and possible neuromas will be documented (presence, location, numbers and (unavoidable) micronerve transections) on a standard map and by digital photomicrography in both groups. The first aim is to confirm their presence and their proximity to the DD fibrosis tissue. Secondly, these allocations will be statistically correlated with clinical outcome and compared between the 2 groups. The ultimate goal of these mappings is to develop new surgical techniques that avoid cutting there nerves and/or cut them at preferable locations (away from recurrence, most likely more proximal at a distance to the proximal interphalangeal joints). Hereby an improved surgical technique (microfasciectomy) can possible reduce/avoid neuroma formation, pain and possibly recurrence.

Also, the presence of nerve growth factor (NGF) will be evaluated. The purpose is to provide information on potential neuro-induced fibrosis. NGF is a cell signalling cytokine that was demonstrated earlier to be associated with nerve tissue, neuromas and pain level. It is linked to the alpha-smooth actin expressing myofibroblast, 'activated' connective tissue cells with contractile properties producing collagen strands that cause the finger contractures. Therefore, the presence of NGF and myofibroblast cells crowd around NGF foci will be studied in a biopsy taken per-operatively. Focus will be on the direct environment of the neuromas. The presence of NGF will also be quantified and compared between both groups. It there is a higher amount of NGF in recurrence, there is a possible role for neuro-induced fibrosis and this creates opportunities to select this protein as a target of treatment to improve clinical outcome.

ELIGIBILITY:
Inclusion criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. The participant or his/her legally authorized representative voluntary signed the informed consent prior to the first assessment
2. Participants are ≥ 18 years and diagnosed with primary/recurrent Dupuytren disease
3. Included patients are eligible for microfasciectomy

Exclusion criteria:

Participants eligible for this study must not meet any of the following criteria:

1. Patients < 18 years
2. Patient included in an interventional trial with an investigational medicinal product
3. Patients with cognitive impairments, severe rheumatic disease and neurological disorders leading to flexion deformities of the fingers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old that present with Dupuytren disease (primary or recurrence) and that are selected for surgery and will undergo the resection of Dupuytren tissue with the microfasciectomy technique.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence of neuromas, NGF, αSMA and S100 | During surgery/microfasciectomy
  Presence of neuromas, NGF, αSMA and S100 in Dupuytren nodules after resection.

SECONDARY OUTCOMES:
Presence of micronerves | During surgery/microfasciectomy
  The presence of micronerves with micro-anatomical description in the digital palmar fascia and their relation to the Dupuytren tissue.
Correlate clinical outcome (motion, pain, recurrence) with these findings (micronerve dissection, presence of neuromas, NGF and αSMA) in both groups | pre-operative, post-operative (10 days, 3 months, 12 months)
  * Objective clinical outcome:
    * Range of motion (by goniometry of Distal interphalangeal, Proximal Interphalangeal and metacarpophalangeal joints)
    * Abe. diathesis scoring
  * Patient reported outcome:
    * QUICK Dash for functionality
    * Visual Analogue Scale (VAS) questionnaire on satisfaction
    * Visual Analogue Scale (VAS) questionnaire on pain

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No